CLINICAL TRIAL: NCT00018187
Title: Combinations of Pharmacologic Smoking Cessation Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADRD-011-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Smoking
Keywords: smoking cessation; bupropion; mecamylamine; nicotine
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Bupropion; Mecamylamine; Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: Bupropion
Drug: Mecamylamine
Drug: Nicotine Patch

SUMMARY:
The purpose of this study is to test the effectiveness of a combination of the drugs bupropion and mecamylamine along with a nicotine patch as a therapy for smoking cessation.

ELIGIBILITY:
Subjects must be a smoker between 20 and 40 years old, have smoked at least 20 cigarettes per day for at least 2 years, wish to stop smoking and be in good general health

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-11; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hartman, M.D.
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States